CLINICAL TRIAL: NCT04281563
Title: The Effect of Medium-chain Triglyceride Oil Massage on Physical Growth in Preterm Infants Weighing Between 1500 and 2000 g: a Prospective Randomized Trial
Brief Title: Medium-chain Triglyceride Oil Massage on Growth in Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 106041
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Preterm Infants; MCT Oil Massage; Growth
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Data were analyzed by a researcher who was not informed of the intervention group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the MCT oil massage (Experimental): The neonates received massage with MCT oil. The 10-min massage intervention consisted of two 5-min phases: tactile and kinesthetic stimulation, which were given three times a day for 7 consecutive days.
  Interventions: Other: massage with MCT oil (group 1)
- massage alone (Placebo Comparator): The neonates received massage without MCT oil. The 10-min massage intervention consisted of two 5-min phases: tactile and kinesthetic stimulation, which were given three times a day for 7 consecutive days.
  Interventions: Other: massage with MCT oil (group 1)
- no massage groups (No Intervention): no intervention

INTERVENTIONS:
Other: massage with MCT oil (group 1) — Two trained nurse took turns performing standardized massage techniques in group 1 and group 2. The difference was that in group 1, the neonates received massage with MCT oil, and in group 2, the neonates received massage without using the oil. The 10-min massage intervention consisted of two 5-min phases: tactile and kinesthetic stimulation (13), which were given three times a day for 7 consecutive days. The massage force was approximately 300 grams, and the massager practiced applying the pressure by using a food scale. The massage was given in the prone and supine positions, and the actions included gentle touching of the head, back and limbs for five 1-min periods, followed by six passive flexion/extension movements lasting 10 s apiece for each arm, then each leg, and finally both legs together for a total of five 1-min periods. Premature infants in the oil massage group received massage with 10 mL/kg/day of MCT oil divided equally into three applications.
  Other Names: massage without MCT oil (group 2)
  Arms: massage alone; the MCT oil massage

SUMMARY:
Aim: To explore the effect of medium-chain triglyceride (MCT) oil massage on growth in preterm infants.

Methods: This randomized controlled trial was conducted in the newborn center of a regional hospital in Taiwan. Preterm infants weighing between 1500 and 2000 g were recruited and randomly assigned to three groups: the MCT oil massage, massage alone and no massage groups. The massages were given three times per day for 7 consecutive days. Weight, length and head circumference were measured in the three groups at birth and on study days 1 to 7.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age between 28 and 37 weeks;
2. weight between 1500 and 2000 g after enrollment;
3. medically stable condition;
4. ≥120 cc per day feeding.

Exclusion Criteria:

1. congenital anomalies;
2. skin disease;
3. requirement for mechanical ventilation;
4. requirement for O2 therapy;
5. presence of fracture.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
weight | on study days 1 to 7
  weight increase

SECONDARY OUTCOMES:
height and head circumference | on study days 1 to 7
  height and head circumference increase

CONTACTS AND LOCATIONS:
Locations (1):
- Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao YC, Wan YH, Chen PH, Hsieh LY. Efficacy of medium-chain triglyceride oil massage on growth in preterm infants: a randomized controlled trial: A CONSORT-compliant article. Medicine (Baltimore). 2021 Jul 30;100(30):e26794. doi: 10.1097/MD.0000000000026794. PMID 34397733